CLINICAL TRIAL: NCT02850315
Title: Assessment Of Intracoronary Thrombus By Optical Frequency Domain Imaging During Percutaneous Coronary Intervention After Successful Fibrinolysis And Its Impact On Myocardial Reperfusion
Brief Title: Intracoronary Thrombus Assessed by OFDI After Successful Fibrinolysis And Its Impact On Myocardial Reperfusion
Acronym: AODIS
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 15-032
Record Dates: First submitted 2016-07-12; First posted 2016-08-01 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-01

CONDITIONS: Myocardial Infarction; Intracoronary Thrombus
Keywords: optimal coherence tomography; myocardial reperfusion
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

INTERVENTIONS:
Device: optimal coherence tomography

SUMMARY:
The pharmacoinvasive approach after thrombolysis is the standard treatment of myocardial infarction when deadlines are too long for primary angioplasty. Coronary angioplasty is then carried out within 3 to 24 hours following thrombolysis. The adjuvant antiplatelet therapy of thrombolysis combines aspirin with clopidogrel (75 or 300 mg depending on age). These clopidogrel doses are associated with a very low anti-platelet aggregation response within 24 hours following administration. However, the antiplatelet agregation that inhibits the progression of intracoronary thrombus must be optimal at the time of angioplasty to reduce the risk of thrombotic events. Intracoronary thrombus residual angiographic post-thrombolysis was associated with impaired myocardial reperfusion but coronary angiography has a very low sensitivity for detecting the thrombus. The optical coherence tomography (OCT) is currently the method of choice to visualize and quantify the intracoronary thrombus. It is used routinely in the presence of a thrombus to correctly estimate the size of the artery and for the evaluation of good stent apposition.

The thrombectomy at the time of angioplasty improves myocardial reperfusion, particularly in case of major thrombotic mass. Intracoronary thrombus residual post-thrombolysis could be a marker for the quality of reperfusion itself correlated to the quality of the antiplatelet post-thrombolysis.

The investigators therefore hypothesize that the systematic use of the OCT before elective angioplasty (within 3 to 24 hours) after successful thrombolysis could be used to guide the use of thrombectomy and adequate stenting and thus improve myocardial reperfusion. Our study will also correlate the importance of the residual thrombus before angioplasty myocardial reperfusion one hand and to the inhibition of platelet activity observed other.

ELIGIBILITY:
Inclusion Criteria:

* acute myocardial infarction
* treated with successful fibrinolysis
* who require coronary stenting

Exclusion Criteria:

* cardiogenic shock
* hemostasis disorders
* non accessible coronary lesion for OCT
* severe renal insuffisiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with acute myocardial infarction treated by successful fibrininolysis and who requires a coronary stenting
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
myocardial reperfusion of systematic guidance measured by OCT of the angioplasty procedure | baseline
  in patients treated with thrombolysis and requiring the establishment of a stent

SECONDARY OUTCOMES:
volume of thrombus messured by OCT before angioplasty | 24hours
inhibition of platelet activity evaluated by aggregometry | 24hours

CONTACTS AND LOCATIONS:
Locations (1):
- ROULE, Caen, France